CLINICAL TRIAL: NCT04469348
Title: Inflammation, Intracellular Invasion and Colonization of the Nasal Mucosa by Staphylococcus Aureus
Acronym: I3COSa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19CH050; 2020-A00321-38 (Other: ANSM)
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Staphylococcus aureus; ICAM-1; nasal cells; S. aureus; nasal swab
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Healthy volunteers will be included. They will have nasal swab at the inclusion visit to detect contamination of S. Aureus.
  * If contamination of S. Aureus: they will have 12 follow-up visits (1 per month)
  * If no contamination of S. Aureus: their participation stops
  Interventions: Diagnostic Test: nasal swab

INTERVENTIONS:
Diagnostic Test: nasal swab — nasal swab will be performed to analysis biological markers at every visit.

SUMMARY:
An inflammatory state of the nasal cells (very close to keratinocytes) could favour the internalization of Staphylococcus aureus and thus constitute a persistent reservoir for the carriage of this bacterium.

Staphylococcus aureus is a commensal bacterium of the skin and mucous membranes that colonizes approximately 2 billion people worldwide Staphylococcus aureus is also a leading cause of community and healthcare-associated infection. Staphylococcus aureus has demonstrated its ability to invade many non-professional phagocytic cell lines such as keratinocytes, osteoblasts, fibroblasts, epithelial cells and endothelial cells. During pro-inflammatory stimulation, internalization of Staphylococcus aureus into keratinocytes is mainly mediated by ICAM-1. These results suggest that, in humans, an inflammatory state of the nasal cells (very close to keratinocytes) could promote the internalization of Staphylococcus aureus and thus constitute a persistent reservoir for the carriage of this bacterium.

DETAILED DESCRIPTION:
The main objective is to compare the expression level of ICAM-1 in nasal cells with and without the presence of Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

* Subject affiliated to a social security scheme or entitled person
* Subject who received informed information about the study et signed consent
* Adult subject (≥18ans)
* Healthy Volunteer

Exclusion Criteria:

* Subject undergoing antibiotic treatment or having received antibiotic treatment (oral, IV or local) in the month prior to inclusion
* Subject with a major haemostasis disorder or anticoagulant treatment contraindicated for surgery
* Subject with a pathology increasing the nasal carriage of S. aureus (chronic furunculosis, diabetes, HIV infection, chronic rhinosinusitis)
* Subject under guardianship or trusteeship
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
level of ICAM-1 expression in nasal cells | Months: 0
  Compare the level of ICAM-1 expression in nasal cells with and without the presence of intracellular Staphylococcus aureus

SECONDARY OUTCOMES:
Measurement of the expression of the genes (mRNA dosage) involved in IL-1 beta secretion | Months: 0
  Measure by rt-qPCR technique.
Measurement of the expression of the genes (mRNA dosage) involved in activation of autophagy | Months: 0
  Measure by rt-qPCR technique.
cytokine concentration | Months: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Measure by analysis of nasal swab.
concentration of ICAM-1 in S. Aureus | Months: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Measure by analysis of nasal swab.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Verhoeven, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No